CLINICAL TRIAL: NCT03709888
Title: An Observational Study Efficacy and Safety of Memantine XR (Extended Release) and Pregabalin Combination Therapy in Chemotherapy-Induced Peripheral Neuropathy (CIPN)
Brief Title: Memantine XR and Pregabalin for Chemotherapy-Induced Peripheral Neuropathy
Status: Completed | Type: Observational
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Principal Investigator, Santosh Kesari, Professor and Director, Saint John's Cancer Institute
Other Study IDs: JWCI-17-0101
Record Dates: First submitted 2018-07-10; First posted 2018-10-17 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Observation Group: Subjects will be identified from patients with chemotherapy induced peripheral neuropathy (CIPN) that are planning to be treated with memantine XR-pregabalin combination therapy.Patients who agree to participate will be asked to complete study questionnaires prior to the start of their CIPN treatment and once per week for six weeks during their treatment.
  Interventions: Drug: Memantine XR-pregabalin combination therapy

INTERVENTIONS:
Drug: Memantine XR-pregabalin combination therapy — Pregabalin and memantine XR work in different pathways and are approved by the U.S. Food and Drug Administration for various indications. Both medications have an established safety profile and have demonstrated improvement on neuropathy-related symptoms.
  Other Names: Namenda XR-Lyrica

SUMMARY:
Study is designed to assess the efficacy and safety of memantine XR and pregabalin in reducing neuropathic pain in patients with chemotherapy-induced peripheral neuropathy (CIPN) caused by prior treatment with any chemotherapy as measured by the Brief Pain Inventory- Short Form (BPI-SF). It will also determine the influence of these drugs on peripheral neuropathy-related functional status and quality of life (QOL) as measured by the EORTC QLQ-C30.

DETAILED DESCRIPTION:
Using an observational, case-only, prospective design, potential subjects will be identified from patients with chemotherapy induced peripheral neuropathy (CIPN) that are planning to be treated with memantine XR-pregabalin combination therapy. The primary objective is to assess the efficacy of memantine XR and pregabalin in reducing neuropathic pain as measured by the Brief Pain Inventory- Short Form (BPI-SF). Patients who agree to participate will be asked to complete study questionnaires prior to the start of their CIPN treatment and once per week for six weeks during their treatment. After this period, patients will be contacted once per month for three months to assess interval medical history, concomitant medications, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

Ability to understand and the willingness to sign a written informed consent. History of any type of cancer treated with chemotherapy.

Chemotherapy induced peripheral neuropathy (CIPN) due to:

* Cisplatin, carboplatin, and oxaliplatin
* Taxanes- paclitaxel, docetaxel, and cabazitaxel
* Thalidomide, lenalidomide, and pomalidomide
* Plant alkaloids, such as vinblastine, vincristine, vinorelbine, and etoposide
* Epothilones, such as ixabepilone
* Bortezomib, carfilzomib
* Eribulin Planning to receive treatment for CIPN with memantine XR and pregabalin. Average daily neuropathic pain intensity > 4 measured by item #5 of BPI-SF (Average daily pain at baseline is the average of pain scores over the last 7 days before enrolling patients in to the study).

CIPN > grade 1 as measured by NCI-CTCAE v 4.0. Must be ≥ 3 months beyond completion of chemotherapy. Not planning to receive concurrent chemotherapeutic agents during the study period.

Patients with diabetes mellitus, peripheral vascular disease, HIV infection, or a significant degenerative or familial neurologic can be included in the study provided they don't have peripheral neuropathy secondary to above mentioned diseases.

Allowable types and amount of prior therapy for neuropathy:

* Patients receiving analgesics for pain associated with CIPN are eligible provided they have taken the same dosage and same medication for at least 2 weeks prior to the study initiation.
* Patients on antidepressants regimens of Selective Serotonin Reuptake Inhibitors (SSRI) or Selective serotonin norepinephrine reuptake inhibitors (SSNRI) for treatment of anxiety or depression, anticonvulsants or mexiletine for the treatment of pain are eligible provided they are on stable dose for 30 days.

Age ≥ 18 years. Both men and women of all races and ethnic groups are eligible for this trial.

Exclusion Criteria:

Any pain other than neuropathic pain of equal or greater severity. Patients with sensory polyneuropathy due to AIDS/HIV, complex regional pain syndrome, and Trigeminal neuralgia.

History of suicidal ideation. Patients with a history of non-compliance. Patients who are judged by the investigator to be unable or unlikely to understand the nature, scope, and possible consequences of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chemotherapy induced peripheral neuropathy (CIPN) that are planning to be treated with memantine XR-pregabalin combination therapy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-07-09 (Actual); Primary Completion 2021-04-29 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Change in average daily pain intensity as measured by the Brief Pain Inventory- Short Form (BPI-SF) | 6 weeks
  Absolute change in the average daily pain intensity as measured by the Brief Pain Inventory- Short Form (BPI-SF) from baseline to the end of 6 weeks measured by item # 5 of Brief Pain Inventory Score (BPI-SF). The BPI assesses pain at its "worst," "least," "average," and "now" (current pain). In clinical trials, the items "worst" and "average" have each been used singly to represent pain severity. A composite of the four pain items (a mean severity score) is sometimes presented as supplemental information.

SECONDARY OUTCOMES:
Change in quality of life (QOL) as measured by European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC QLQ-C30) | 6 weeks
  Absolute change in the QoL measured by European Organisation for Research and Treatment of Cancer Quality-of-life Questionnaire Core 30 (EORTC QLQ-C30) after 6 weeks of treatment compared to baseline. The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items. Each of the multi-item scales includes a different set of items - no item occurs in more than one scale. All of the scales and single-item measures range in score from 0 to 100. A high scale score represents a higher response level.
Change in the intensity of mechanical allodynia measured using qualitative sensory testing | 6 weeks
  Absolute change in mechanical allodynia intensity after 6 weeks of treatment compared to baseline. Testing is done by touching the sensitive (neuropathic) area with a foam brush 3 times in 5 secs and asking the patient about their pain score before and after the procedure.
Change in neuropathic symptoms as measured by Neuropathic Pain Symptom Inventory (NPSI) | 6 weeks
  Absolute change in neuropathic symptoms measured by Neuropathic Pain Symptom Inventory (NPSI) scores after 6 weeks of treatment compared to baseline. A total intensity score can be calculated as the sum of the scores of the 10 descriptors ranging from 0 to 100. Five subscores corresponding to the mean scores of the items belonging to each of the five dimensions ranging from 0 to 10. ) is "no pain" and 10 is "the most intense pain imaginable".
Change in reported sleep interference as measured by item # 9 of Brief Pain Inventory- Short Form (BPI-SF) | 6 weeks
  Absolute change in sleep interference measured by item # 9 of Brief Pain Inventory Score (BPI-SF) after 6 weeks of treatment from baseline. Score for question 9F for sleep ranges from 0 "does not interfere" to 10 "completely interferes".

CONTACTS AND LOCATIONS:
Overall Officials: Santosh Kesari, MD, PhD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- John Wayne Cancer Institute at Providence Saint John's Health Center, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided